CLINICAL TRIAL: NCT06307288
Title: Efficacy and Safety of Tranilast Combined With Minocycline in the Treatment of Rosacea
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240301-2
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Rosacea
Keywords: rosacea; mast cell stabilizers; tranilast; minocycline; treatment; clinical research
MeSH Terms: conditions — Rosacea; cyclopia sequence | interventions — Minocycline; tranilast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- minocycline treatment group (Experimental): The patient was treated with oral minocycline capsules, 50mg each time, once a day, for 12 weeks.
  Interventions: Drug: minocycline
- tranilast treatment group (Experimental): The patient was treated with oral tranilast capsules, 0.1g each time, three times a day, for 12 weeks.
  Interventions: Drug: tranilast
- tranilast combined with minocycline treatment group (Experimental): The patient was treated with oral tranilast capsules, 0.1g each time, three times a day; oral minocycline capsules, 50mg each time, once a day, for 12 weeks.
  Interventions: Drug: minocycline; Drug: tranilast

INTERVENTIONS:
Drug: minocycline — The patient was treated with oral minocycline, 50mg each time, once a day, for 12 weeks.
  Arms: minocycline treatment group; tranilast combined with minocycline treatment group
Drug: tranilast — The patient was treated with oral tranilast, 0.1g each time, three times a day, for 12 weeks.
  Arms: tranilast combined with minocycline treatment group; tranilast treatment group

SUMMARY:
Rosacea is a chronic inflammatory skin disease with a complex pathogenesis involving multiple factors. Currently, the treatment of rosacea remains highly challenging. Mast cells, as key participants in the pathogenesis of rosacea, have been shown to alleviate rosacea symptoms with some topical, oral, and injectable mast cell stabilizers in recent years. Tranilast stabilizes mast cells and basophils by acting on their cell membranes and preventing their degranulation. Tranilast has been used in the treatment of various skin disease, such as hypertrophic scars and atopic dermatitis. Minocycline is a first-line treatment for rosacea, and low-dose minocycline treatment (50mg/day) is believed to have anti-inflammatory effects without antibacterial effects, thus minimizing the dysbiosis and bacterial resistance caused by antibiotic use. Therefore, this study aims to investigate the effectiveness and safety of combining mast cell stabilizer tranilast with low-dose minocycline treatment for rosacea, providing new treatment options and insights for rosacea patients.

DETAILED DESCRIPTION:
Rosacea is a chronic inflammatory skin disease with a complex pathogenesis involving multiple factors. Currently, the treatment of rosacea remains highly challenging. In the skin, mast cells are located in the dermis near nerve endings and blood vessels, playing a crucial role in inflammatory responses. Mast cells, as key participants in the pathogenesis of rosacea, have been shown to alleviate rosacea symptoms with some topical, oral, and injectable mast cell stabilizers in recent years. Tranilast stabilizes mast cells and basophils by acting on their cell membranes and preventing their degranulation. Tranilast has been used in the treatment of various skin disease, such as hypertrophic scars and atopic dermatitis. Minocycline is a first-line treatment for rosacea, and low-dose minocycline treatment (50mg/day) is believed to have anti-inflammatory effects without antibacterial effects, thus minimizing the dysbiosis and bacterial resistance caused by antibiotic use. However, there is currently a lack of clinical studies evaluating the efficacy and safety of combined treatment with tranilast and minocycline for rosacea. Therefore, this study aims to investigate the effectiveness and safety of combining mast cell stabilizer tranilast with low-dose minocycline treatment for rosacea, providing new treatment options and insights for rosacea patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females, aged 18-60 years old;
2. Diagnosed with erythematotelangiectatic or papulopustular rosacea, with an investigator' s global assessment of 3-5;
3. Patients with good cognitive function and normal mental status;
4. Patients with good communication skills;
5. Voluntary participation in the study and signing of informed consent form.

Exclusion Criteria:

1. Allergy to any component of tranilast capsules;
2. Allergy to any component of minocycline capsules;
3. History of systemic medication for rosacea treatment within the past month;
4. Pregnancy or lactation;
5. Presence of severe primary diseases in addition to rosacea, such as cardiovascular system, cerebrovascular system, digestive system, urinary system, hematopoietic system diseases, or systemic failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
lesion counts | From enrollment to week 12
  The counts of skin lesions, including papules, pustules, and papulopustules, was used to evaluate the changes of facial inflammatory skin lesions before and after treatment.
Clinician's Erythema Assessment score | From enrollment to week 12
  The name of the scale is Clinician's Erythema Assessment. It was used to evaluate the change of persistent facial erythema before and after treatment. The score on the Clinician's Erythema Assessment scale ranges from 0 to 9, with higher scores indicating more severe persistent erythema on the patient's face.
Global Flushing Severity Scale score | From enrollment to week 12
  The name of the scale is Global Flushing Severity Scale. It was used to evaluate the change of facial flushing symptoms before and after treatment. The score on the Global Flushing Severity Scale ranges from 0 to 10, with higher scores indicating more severe symptoms of facial flushing.
Global Acne Grading System score | From enrollment to week 12
  The name of the scale is Global Acne Grading System. It was used to evaluate the changes of facial inflammatory skin lesions before and after treatment. The Global Acne Grading System score ranges from 0 to 32, with higher scores indicating more inflammatory lesions on the patient's face.

SECONDARY OUTCOMES:
patient satisfaction evaluation | week 12
  Patient satisfaction was evaluated as very satisfied, satisfied, relatively satisfied and dissatisfied.
melanin index | From enrollment to week 12
  Use non-invasive skin analyzer to measure the melanin index on the patient's facial skin at each follow-up visit.
erythema index | From enrollment to week 12
  Use non-invasive skin analyzer to measure the erythema index on the patient's facial skin at each follow-up visit.
transepidermal water loss | From enrollment to week 12
  Use non-invasive skin analyzer to measure the transepidermal water loss on the patient's facial skin at each follow-up visit.
Dermatology Life Quality Index score | week 0 and12
  The name of the scale is Dermatology Life Quality Index. It was used to assess the changes in quality of life before and after treatment. The Dermatology Life Quality Index score ranges from 0 to 29, with higher scores indicating a greater impact of the disease on the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong Universi, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marchitto MC, Chien AL. Mast Cell Stabilizers in the Treatment of Rosacea: A Review of Existing and Emerging Therapies. Dermatol Ther (Heidelb). 2021 Oct;11(5):1541-1549. doi: 10.1007/s13555-021-00597-7. Epub 2021 Sep 2. PMID 34476755
- [Result] Aroni K, Tsagroni E, Kavantzas N, Patsouris E, Ioannidis E. A study of the pathogenesis of rosacea: how angiogenesis and mast cells may participate in a complex multifactorial process. Arch Dermatol Res. 2008 Mar;300(3):125-31. doi: 10.1007/s00403-007-0816-z. Epub 2007 Dec 11. PMID 18071725
- [Result] Wozniak E, Owczarczyk-Saczonek A, Lange M, Czarny J, Wygonowska E, Placek W, Nedoszytko B. The Role of Mast Cells in the Induction and Maintenance of Inflammation in Selected Skin Diseases. Int J Mol Sci. 2023 Apr 10;24(8):7021. doi: 10.3390/ijms24087021. PMID 37108184
- [Result] Del Rosso JQ, Webster G, Weiss JS, Bhatia ND, Gold LS, Kircik L. Nonantibiotic Properties of Tetracyclines in Rosacea and Their Clinical Implications. J Clin Aesthet Dermatol. 2021 Aug;14(8):14-21. Epub 2021 Aug 1. PMID 34840653
- [Result] Schaller M, Almeida LMC, Bewley A, Cribier B, Del Rosso J, Dlova NC, Gallo RL, Granstein RD, Kautz G, Mannis MJ, Micali G, Oon HH, Rajagopalan M, Steinhoff M, Tanghetti E, Thiboutot D, Troielli P, Webster G, Zierhut M, van Zuuren EJ, Tan J. Recommendations for rosacea diagnosis, classification and management: update from the global ROSacea COnsensus 2019 panel. Br J Dermatol. 2020 May;182(5):1269-1276. doi: 10.1111/bjd.18420. Epub 2019 Oct 16. PMID 31392722
- [Result] Tan J, Almeida LM, Bewley A, Cribier B, Dlova NC, Gallo R, Kautz G, Mannis M, Oon HH, Rajagopalan M, Steinhoff M, Thiboutot D, Troielli P, Webster G, Wu Y, van Zuuren EJ, Schaller M. Updating the diagnosis, classification and assessment of rosacea: recommendations from the global ROSacea COnsensus (ROSCO) panel. Br J Dermatol. 2017 Feb;176(2):431-438. doi: 10.1111/bjd.15122. Epub 2017 Jan 23. PMID 27718519
- [Result] Schaller M, Almeida LM, Bewley A, Cribier B, Dlova NC, Kautz G, Mannis M, Oon HH, Rajagopalan M, Steinhoff M, Thiboutot D, Troielli P, Webster G, Wu Y, van Zuuren E, Tan J. Rosacea treatment update: recommendations from the global ROSacea COnsensus (ROSCO) panel. Br J Dermatol. 2017 Feb;176(2):465-471. doi: 10.1111/bjd.15173. Epub 2017 Feb 5. PMID 27861741